CLINICAL TRIAL: NCT01003678
Title: A Phase I Study Evaluating the Safety and Tolerability of Oral Clofarabine in Intermediate to High Risk Myelodysplastic Patients
Brief Title: Safety and Tolerability of Oral Clofarabine in Intermediate to High Risk Myelodysplastic Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug provider withdrew support
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 144208
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic syndrome; Clofarabine; low-dose oral clofarabine; intermediate risk Myelodysplastic syndrome; high risk Myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Level 1 (Experimental): 1 mg daily for 5 consecutive days followed by 23 days off drug
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Dose Escalation Schedule - Level 1: 1 mg daily x 5 days (orally) followed by 23 days off drug.
  Levels 2, 3, 4 and 5 are: 3, 5, 10 and 15 mg daily x 5 days followed by 23 days off drug.

SUMMARY:
This is a Phase I trial for patients with intermediate or high risk myelodysplastic syndrome (MDS).

The study agent, clofarabine, is produced by Genzyme Pharmaceuticals.

DETAILED DESCRIPTION:
The specific purpose of the study is to determine the safety, maximum tolerated dose (MTD) and recommended Phase II dose of clofarabine in patients with MDS.

* We will start at a dose of 1 mg daily.
* We will treat a group of 3 patients with clofarabine at that dose level.
* If there are no severe side effects seen at that dose level, then the next group of 3 patients will receive a higher dose.
* Treatment of groups of 3 patients will continue at higher dose levels until severe side-effects are noted.
* If more than 1 of the 3 patients experiences a severe side effect, dosing will be stopped at that level.
* If only one of the three patients experience a severe side effect, then three more patients will be treated, at that dose level and if they too experience severe side effects, then dose escalation will be stopped and the maximum tolerated dose will be determined.
* 10 more patients will be enrolled at the maximum tolerated dose.
* There will be up to 5 dose levels tested.
* We plan to test how much of the drugs are in the patient's blood at different times, and the levels of certain proteins in their blood.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent.
* Patients with MDS must have IPSS score that falls in the intermediate or high risk disease (intermediate 1 will have to be transfusion dependent).
* Patients may have received up to two prior therapies for MDS including one hypomethylating agent and/or a biologic agent (biologic agents include GM-CSF or equivalent, danazol or equivalent, Sunitinib, Revlimid, ATG, or a vaccine).
* Age ≥ 18
* Have adequate renal and hepatic functions as indicated by the following laboratory values:

  * Serum creatinine ≤ 1 mg/dL; if serum creatinine >l mg/dL, then the estimated glomerular filtration rate (GFR) must be >50 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation.
  * Serum bilirubin ≤1.5 mg/dL x upper limit of normal (ULN)
  * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤2.5 x ULN
  * Alkaline phosphatase ≤2.5 x ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Active CNS disease
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Have had any prior treatment with clofarabine
* Have had a diagnosis of another malignancy, unless the patient has been disease free for at least 3 years following the completion of curative intent therapy, with the following exceptions:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
* Have prior positive test for the Human Immunodeficiency Virus (HN).
* Have prior positive test for the Human Immunodeficiency Virus (HN).
* Have currently active gastrointestinal disease, or prior surgery that may affect the ability of the patient to absorb oral clofarabine.
* Patients taking proton pump inhibitors such as omeprazole (Prilosec®), lansoprazole (Prevacid®), or esomeprazole (Nexium®). Those who cannot stop taking these drugs should be switched to H2 blockers such as famotidine (Pepcid®)or ranitidine (Zantac®).
* Patients taking alternative medicines (such as herbal or botanical) are not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety, maximum tolerated dose (MTD) and recommended phase II dose of Clofarabine in patients with myelodysplastic syndrome (MDS). | Up to 6 months

SECONDARY OUTCOMES:
To determine the efficacy of Clofarabine in patients with MDS | Up to 6 months
To determine the differences in clofarabine triphosphate levels in cells following clofarabine treatment | Pre, Day 1: Hourly for 6 hours, Pre Day 5:Hourly for 5 hours
Determine the differences in clofarabine plasma levels following clofarabine treatment | Pre, Day 1: Hourly for 6 hours, Pre Day 5:Hourly for 5 hours
Evaluate the effect of clofarabine on DNA methylation | Pre and Day 1
Estimate post-treatment p53R2levels in patients treated at the MTD (in the expanded cohort) | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wetzler Meir, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States